CLINICAL TRIAL: NCT03485196
Title: The Relationship Between Microsatellite Instability and Efficacy of Fluorouracil Based Adjuvant Chemotherapy in Gastric Cancer After Operation
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Qinghai University (Other)
Collaborators: Qinghai People's Hospital (Other); LanZhou University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Other Study IDs: AHQU-2017003
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
Keywords: Microsatellite Instability; Fluorouracil; Adjuvant chemotherapy; Efficacy; Operation
MeSH Terms: conditions — Stomach Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MSI-H group: We use the immunohistochemical expression of mismatch repair proteins (MutS protein homolog 2( MSH2),MutS protein homolog 6( MSH6) and PMS2（postmeiotic segregation increased 2 ）) to Determine the MSI status . When one antibodies or more show negative nuclear staining of the tumor cells, the MSI state can be defined as Microsatellite instability high (MSI-H).
  Interventions: Other: Microsatellite instability
- MSI-L group: We use the immunohistochemical expression of mismatch repair proteins (MLH1, MSH2, MSH6 and PMS2) to Determine the MSI status . when all the four antibodies show positive nuclear staining of the tumor cells, the MSI state can be defined as Microsatellite stable (MSI-L).
  Interventions: Other: Microsatellite instability
- MSS group: We use the immunohistochemical expression of mismatch repair proteins (MLH1, MSH2, MSH6 and PMS2) to Determine the MSI status . when all the four antibodies show positive nuclear staining of the tumor cells, the MSI state can be defined as Microsatellite stable (MSS).
  Interventions: Other: Microsatellite instability

INTERVENTIONS:
Other: Microsatellite instability — The microsatellite instability status are definite to three type:MSI-H, MSI-L,and MSS. The gastric cancer patients who received D2 resection were included in 3 groups：MSI-H group， MSI-L group，and MSS group. All patient must be accept fluorouracil(5-FU) based adjuvant chemotherapy. We will analyze the relationship between MSI status and efficacy of 5-FU based adjuvant chemotherapy by observing the survival period of patients with different MSI status.

SUMMARY:
The relationship between Microsatellite instability and efficacy of fluorouracil based adjuvant chemotherapy in gastric cancer after operation.

DETAILED DESCRIPTION:
To explore the relationship between Microsatellite instability and efficacy of fluorouracil based adjuvant chemotherapy in gastric cancer after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology or cytopathology proven gastric cancer;
2. Operable advanced gastric cancer patients: primary lesions can be completely excision, no distant metastasis;
3. Postoperative patients who can tolerate 5-FU based (5-FU，S-1 or Capecitabine) adjuvant chemotherapy;
4. Life expectancy of at least 6 months;
5. ECOG（Eastern Cooperative Oncology Group ） score 0-1;
6. Age: 18~80 years old;
7. Normal hemodynamic indices before the recruitment (including blood cell count and liver/kidney function).

   * For example: WBC（White blood cell count ）>4.0×109/L; NEU（Neutrophils）>1.5×109/L; PLT（Platelet）>100×109/L;
8. Roughly normal cardiopulmonary function: No coronary heart disease, myocardial infarction, pulmonary heart disease, refractory hypertension;
9. Not concomitant with other uncontrollable benign diseases before the recruitment;

9. Voluntarily signed the informed consent.

Exclusion Criteria:

1. Advanced gastric cancer patients with distant metastasis and inoperable ;
2. Patients who cannot tolerate 5-FU based adjuvant chemotherapy;
3. Pregnant or lactating women;
4. Patients who have no desire to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  The time from the primary operation to disease recurrence or death.

SECONDARY OUTCOMES:
Overall survival(OS) | 5 years
  The The time from operation to death or the last follow-up. The time from operation to death or the last follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Second Hospital Affiliated to Lanzhou University, Lanzhou, Gansu
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - People's Hospital of Qinghai Province, Xining, Qinghai

IPD SHARING:
Plan to Share IPD: No